CLINICAL TRIAL: NCT03823040
Title: Oxiconazole Nitrate Solid Lipid Nanoparticles : Formulation, In-vitro Characterization and Clinical Assessment of An Analogous Loaded Carbopol Gel
Brief Title: Clinical Assessment of Oxiconazole Nitrate Solid Lipid Nanoparticles Loaded Gel
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Heba Mansour, Assistant professor of pharmaceutics, Faculty of Pharmacy, Minia University, Minia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: OXIHebaSLNs
Record Dates: First submitted 2019-01-19; First posted 2019-01-30 (Actual); Last update posted 2019-01-30 (Actual); Status verified 2019-01

CONDITIONS: Tinea
MeSH Terms: conditions — Tinea

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tinox® group (Active Comparator): Male patients (12 to 43 years old) including 5 cases tinea pedis, 9 tinea versicolor and treated with oxiconazole nitrate cream 1%.
  Interventions: Drug: Oxiconazole Nitrate Cream 1%
- Oxiconazole nitrate SLNs loaded gel group (Experimental): 13 males and one female (17 to 50 years old) including 3 cases tinea pedis, 8 tinea versicolor, 3 tinea circinate and treated with oxiconazole nitrate SLNs loaded gel
  Interventions: Drug: Oxiconazole nitrate SLNs loaded gel.

INTERVENTIONS:
Drug: Oxiconazole Nitrate Cream 1% — Tinox® group was treated with oxiconazole nitrate cream 1 % . Treatment was performed by rubbing the cream twice daily for two/ four weeks according to different types of tinea.
  Other Names: Tinox® cream 1 %
  Arms: Tinox® group
Drug: Oxiconazole nitrate SLNs loaded gel. — Oxiconazole nitrate SLNs loaded gel group was treated with oxiconazole nitrate SLNs loaded gel.Treatment was performed by rubbing the gel twice daily for two/ four weeks according to different types of tinea.
  Other Names: Developed SLNs gel
  Arms: Oxiconazole nitrate SLNs loaded gel group

SUMMARY:
Clinical study for the developed oxiconazole nitrate solid lipid nanoparticles (SLNs) gel system compared to the corresponding marketed product was conducted on 28 patients with different types of tinea fungal infection.

DETAILED DESCRIPTION:
The clinical work has been carried out in accordance with The Code of Ethics of the World Medical Association for experiments involving humans. The study was conducted on 28 patients (12 to 50 years old) with tinea of different types attending the dermatology department outpatient clinic of Minia University Hospital. Local institutional review board approval was obtained for this study (ethical approval number is 23/12). Pregnant females and patients with Immunocompromising disease,open wounds and psychological disorders were excluded. Patients were subjected to skin irritation test by applying gel on an area of 2 square inch to the back of hand. Then, examination for the presence of lesion or irritation was conducted. The patients divided into two groups of 14 patients each. Tinox® group was male patients from 12 to 43 years old. The included cases were 5 tinea pedis, 9 tinea versicolor. Oxiconazole nitrate SLNs loaded gel group was 13 males and one female from17 to 50 years old. The included cases were 3 tinea pedis, 8 tinea versicolor, 3 tinea circinate. An informed consent has been obtained from all patients enrolled in the study for photography and treatment. History, general local examination and laboratory investigation for all patients were conducted.The patients were clinically examined after determining the type of infection. Tinox® group was treated with Tinox® cream 1 % while oxiconazole nitrate SLNs loaded gel group was treated with the oxiconazole nitrate SLNs-loaded gel. Treatment was performed by rubbing the cream or gel twice daily for two/ four weeks according to different types of tinea. Patients were advised to avoid sun exposure between 10 am and 4 pm and avoid removal of the applied dose during the period of follow up, the clinical improvement of the patients and length of treatment was assessed according to quartile grading scale patient satisfaction. It was rated by the patient and the physician as excellent, good, fair and poor according to the following criteria. Excellent: both the patient and the physician agreed that the result was satisfactory. Good: the result although acceptable was not quite up to expectation of the patient, but the physicians were pleased with the outcome. Fair: the improvement was evaluated by both the patient and the physician to be less than expected but still with same improvement. Poor: unsatisfactory results to the patient and /or the physician. All adverse effects were checked during study.High resolution digital photographs were taken for lesions of all patients using identical camera folder setting before starting and one-month post treatment. Clinical improvement was evaluated by physicians through comparing photographs. The criteria for evaluations using a quartile grading scale was: 0=no improvement. 1=mild (percent improvement, less than 25%), 2=moderate (percent improvement 25-49%), 3=good (percent improvement 50-74%), 4=excellent (percent improvement more than 75%). In addition, a patient satisfaction score was rated using the following scale, A. not satisfied, B. somewhat satisfied, C. highly satisfied.

Skin scrapes were taken from each group before and after treatment. All skin scrapes were routinely processed by potassium hydroxide 20% to be examined for presence of fungal elements. A built-in camera and a light microscope were used to photograph and examine the sectioned skin areas.

IBM SPSS® ( International business machine statistical Package for the Social Sciences (version 22, USA) was utilised for data analysis. The acceptability of the tested formulations was assessed using the chi-square test, P ≤ 0.05 was considered statistically significant. All the results were presented as the mean ± standard deviation (SD).

ELIGIBILITY:
Inclusion Criteria:

* patients with different types of tine infection

Exclusion Criteria:

* Pregnant females and patients with Immunocompromising disease, open wounds and psychological disorders were excluded.

Ages: 12 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 28 (Actual)
Dates: Start 2018-07-16 (Actual); Primary Completion 2018-12-23 (Actual); Study Completion 2018-12-30 (Actual)

PRIMARY OUTCOMES:
Measurement of clinical improvement using quartile grading scale patient satisfaction | one month
  the clinical improvement of the patients was assessed according to quartile grading scale patient satisfaction. It was rated by the patient and the physician as excellent, good, fair and poor according to the following criteria. Excellent: both the patient and the physician agreed that the result was satisfactory. Good: the result although acceptable was not quite up to expectation of the patient, but the physicians were pleased with the outcome. Fair: the improvement was evaluated by both the patient and the physician to be less than expected but still with same improvement. Poor: unsatisfactory results to the patient and /or the physician. All adverse effects were checked during study.

SECONDARY OUTCOMES:
Microscopical examination of skin scrapes for detection of fungal elements | one month
  Skin scrapes were taken from each group before and after treatment. All skin scrapes were routinely processed by potassium hydroxide 20% to be examined for presence of fungal elements. A built-in camera and a light microscope were used to photograph and examine the sectioned skin areas.

CONTACTS AND LOCATIONS:
Overall Officials: Heba F Mansour, Ph.D, Study Director — Associate professor of Pharmaceutics, Faculty of Pharmacy, Minia and Deray University, Minia, Egypt.
Locations (1):
- Minia University Hospital,dermatology department, out patient clinic, Minya, Egypt

IPD SHARING:
Plan to Share IPD: Undecided